CLINICAL TRIAL: NCT01855685
Title: A Phase I/II, Non Randomized, Multicenter, Open-label Study of Autologous CD34+ Cells Transduced With the G1XCGD Lentiviral Vector in Patients With X-linked Chronic Granulomatous Disease
Brief Title: Gene Therapy for X-linked Chronic Granulomatous Disease (X-CGD)
Acronym: CGD
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G1XCGD.01
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: X-Linked Chronic Granulomatous Disease
Keywords: XCGD, lentivirus, cellular therapy
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental): X vivo gene therapy
  Interventions: Genetic: X vivo gene therapy

INTERVENTIONS:
Genetic: X vivo gene therapy — Transplantation of patient's autologous CD34+ cells transduced with lentiviral vector containing GP91PHOX gene

SUMMARY:
X-linked chronic granulomatous disease (X-CGD) is a rare genetic disorder, which affects boys. It is caused by an error in a gene that makes part of the immune system. The basic defect lies in specialised white blood cells called phagocytic cells (or phagocytes), which are responsible for protection against infection by destroying invading bacteria and fungi. They do this by pouring large amounts of substances similar to bleach onto these organisms. In CGD, there is a defect in the system that makes the bleach, called the NADPH-oxidase. In X-CGD (which accounts for two thirds of patients), the defect lies in a gene which makes up a critical part of the NADPH-oxidase (known as gp91-phox), and the cells cannot make bleach-like substances. Therefore they kill bacteria and fungi poorly, and the patients suffer from severe and recurrent infections. This also results in inflammation which can damage parts of the body such as the lung and gut.

In many cases, patients can be adequately protected from infection by constant intake of antibiotics. However, in others, severe life-threatening infections break through. In some cases, inflammation in the bowel or urinary systems results in blockages which cannot be treated with antibiotics, and which may require the use of other drugs such as steroids. Development of curative treatments for CGD is therefore of great importance.

ELIGIBILITY:
Inclusion Criteria:

* Male X-CGD patients
* Molecular diagnosis confirmed by DNA sequencing
* At least one prior ongoing or resistant severe infection and/or inflammatory complications requiring hospitalisation despite conventional therapy
* No HLA-matched donor available after 3 months search unless the risk of waiting for a potential match or for performing an allogeneic transplant is considered unacceptable by the investigator

Exclusion Criteria:

* Contraindication for leukapheresis
* Contraindication for administration of conditioning medication
* Administration of gammainterferon within 30 days before the infusion of transduced autologous CD34+ cells

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Safety of the procedure as measured by the incidence of adverse events | 24 months
Restoration and stability over time of the NADPH functioning granulocytes assessed by a DHR test | 12 months

SECONDARY OUTCOMES:
Normalisation of nutritional status, growth, development, severe infection and/or inflammatory complication which recommended patient's inclusion | 24 months
Percentage of transduced CD34+ haematopoietic cells infused and of blood cells over time | 24 months
Immunological reconstitution | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Thrasher, MD, PHD, Principal Investigator — Great Ormond Street Hospital NHS Foundation Trust - London - UK; Janine Reichenbach, MD, Principal Investigator — University Children's Hospital Zürich - Switzerland; Hubert Serve, MD, PHD, Principal Investigator — Department of Hematology/Oncology, University Hospital Frankfurt and Institute for Biomedical Research, Georg-Speyer-Haus, Frankfurt - Germany; Emma Morris, MD, PHD, Principal Investigator — Royal Free Hospital / University College London Hospital (UCLH)
Locations (2):
- United Kingdom (2):
  - University College London Hospital (UCLH), London
  - Great Ormond Street Hospital NHS Foundation Trust, London